CLINICAL TRIAL: NCT00457223
Title: Randomized Controlled Trial to Compare Fibrin Glue and Suture in Primary Pterygium Excision With Amniotic Membrane Transplantation
Brief Title: To Compare Fibrin Glue and Suture in Primary Pterygium Excision With Amniotic Membrane Transplantation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Ratchadapiseksompotch Fund, Chulalongkorn University, Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 401/49
Record Dates: First submitted 2007-04-04; First posted 2007-04-06 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2008-02

CONDITIONS: Pterygium
Keywords: pterygium; pterygia; excision; amniotic membrane transplantation; fibrin glue; suture
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1Fibrin glue (Experimental): After pterygium excision, amniotic membrane was shaped and attached to bare scleral area using fibrin glue (Quixil®)
  Interventions: Procedure: Amniotic membrane transplantation using fibrin glue
- 2 Suture (Active Comparator): After pterygium excision, amniotic membrane was shaped and attached to bare scleral area using continuous suture with nylon 10-0
  Interventions: Procedure: Amniotic membrane transplantation using fibrin glue

INTERVENTIONS:
Procedure: Amniotic membrane transplantation using fibrin glue — After pterygium excision, amniotic membrane was shaped and attached to bare scleral area using fibrin glue (Quixil®) in 16 eyes of 16 patients of FG group and continuous suture with nylon 10-0 in 16 eyes of 16 patients of SU group.
  Other Names: Quixil®; Nylon 10-0

SUMMARY:
The purpose of this study is to compared between conventional pterygium excision and AMT transplantation with suture and with fibrin glue.

DETAILED DESCRIPTION:
There are few studies about use of fibrin glue in pterygium surgery with conjunctival auto-graft with promising outcome. Less recurrent rate, less discomfort and halve surgical time were reported.

Up to our knowledge,there is no report of fibrin glue in pterygium excision with amniotic membrane transplantation(AMT). There is conventional technique to use AMT in King Chulalongkorn Memorial Hospital because some benefits over conjunctival auto-graft e.g.

* Preserve healthy superior conjunctiva for future glaucoma filtering surgery
* Can use in big or 2-headed pterygium
* Not contract as conjunctival graft esp. in case of fibrin glue
* Potential easier to use with fibrin glue
* Available from Thai Red Cross Eye Bank Comparison(s): amniotic membrane transplantation using fibrin glue compare to suture after pterygium excision.

ELIGIBILITY:
Inclusion Criteria:

* primary pterygium

Exclusion Criteria:

* Pregnant women
* Recurrent pterygium
* Pseudopterygium
* Uncontrolled systemic disease.
* Known allergy to any of the study agents or preservatives used in the formulations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Pain and discomfort during and after surgery using visual analog scale | during surgery and after surgery up to 30 days

SECONDARY OUTCOMES:
Surgical time | start and to the end of surgery
Healing of epithelial defect on cornea and AMT | until 30 days
Postoperative inflammation | up to 30 days
Complications e.g. Recurrent, graft loss/dehiscent, re-operation | until last follow up

CONTACTS AND LOCATIONS:
Overall Officials: Ngamjit Kasetsuwan, MD, Study Chair — Ophthalmology Department, Faculty of Medicine, Chulalongkorn University
Locations (1):
- Department of Ophthalmology, King Chulalongkorn Memorial hospital, Bangkok, Thailand